CLINICAL TRIAL: NCT01075399
Title: A Pilot, Phase II , Open Label, Nonrandomized, Multi- Center Study of [F 18]HX4 Positron Emission Tomography (PET) to Detect Hypoxia in Tumors
Brief Title: Study of [F 18]HX4 Positron Emission Tomography (PET) as a Tool to Detect Hypoxia in Tumors
Acronym: HX4-200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HX4-200
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-07

CONDITIONS: Head and Neck Cancer; Lung Cancer; Liver Cancer; Rectal Cancer; Cervical Cancer
Keywords: [F 18]HX4; HX4; Hypoxia; Head/Neck Cancer; Lung Cancer; Liver Cancer; Rectal Cancer; Cervical Cancer; HIF1 alpha; CAIX
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Liver Neoplasms; Rectal Neoplasms; Uterine Cervical Neoplasms; Hypoxia | interventions — 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F 18]HX4 (Experimental): [F18]HX4, 10 mCi, is administered in a single intravenous bolus injection, followed by a saline flush.
  Interventions: Drug: [F 18]HX4

INTERVENTIONS:
Drug: [F 18]HX4 — Approximately forty (40) patients who have diagnosis confirmed by histopathological examination of tumor tissue from head/neck, lung, liver, rectal or cervical cancers and will receive chemotherapy, radiation therapy or chemoradiotherapy, will be imaged under PET/CT with [F 18]HX4
  Other Names: [F-18]HX4; 3-[18F]fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl); -1H-1,2,3-triazol-1-yl)-propan-1-ol

SUMMARY:
This pilot phase II study is designed as a test and retest study to investigate [F 18]HX4 as a reliable non-invasive PET imaging marker for detection of tumor hypoxia regions and to establish a threshold for [F 18]HX4 uptake in the tumor. The study will evaluate the relationship between hypoxia biomarkers (HIF1α and CA-IX) by immunohistochemistry (IHC) and tumor uptake of [F 18]HX4 by PET imaging.

DETAILED DESCRIPTION:
A Pilot Phase II Study

The primary objectives for this study are:

* To test the reproducibility of [F-18] HX-4 uptake in tumors by imaging the same patient on sequential days in a test-retest protocol
* To test and confirm the relationship between hypoxia in tumors measured by hypoxia related biomarkers (HIF1α and CA-IX) with immunohistochemistry (IHC) and regional [F-18 HX-4] uptake in tumors with PET/CT.

The secondary objectives for this study are:

* To continue safety evaluation by the collection of safety data from all patients
* To establish the threshold for hypoxia uptake in [F- 18]HX4 PET imaging
* To collect data to test [F-18]HX4 PET imaging as a predictor of response in a subgroup of patients receiving treatment
* To gain experience with [F-18]HX4 PET/CT in order to improve the study design to conduct future studies

Design: An open label, non-randomized, uncontrolled, single group assignment, pilot efficacy study

Procedures: Informed consent, collection of demographic information, medical history, blood labs, physical examination, vital signs, ECGs, two or three sets of [F-18]HX4 dosing and imaging scans including two pretreatment, and one mid-treatment if [F-18]HX4 tumor/background ratio ≥ 1.3 from pre-treatment scans, one pre-treatment [F-18]FDG, one mid-treatment if [F- 18]HX4 tumor/background ratio ≥1.3 from pre-treatment scans, concomitant medication collection, adverse event monitoring, and assessment of tumor response to treatment

Patients: Approximately forty (40) patients who have diagnosis confirmed by histopathological examination of tumor tissue from head/neck, lung, liver, rectal or cervical cancers and will receive chemotherapy, radiation therapy or chemoradiotherapy. This allows for approximately 30 evaluable patients to complete this study at approximately six sites.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years and male or female of any race / ethnicity
* Patient or patient's legally acceptable representative provides written informed consent and is willing to comply with protocol procedures
* Patient must have histopathologically confirmed head/neck, lung, liver, rectal or cervical cancer with tumor size ≥ 3cm
* Patient has tumor tissue samples available before treatment for future immunohistochemistry biomarker tests (HIF1alpha and CA-IX)
* Patient is scheduled to have or already had a clinical [F 18]FDG PET/CT scan recommended to be within 14 days of the first pre-treatment [F 18]HX4 PET/CT scan and have no treatment intervention in between these two scans
* Patient is scheduled or is intended to be scheduled to receive chemotherapy, radiation or chemoradiotherapy treatment(s) after the pre-treatment [F 18]HX4 PET/CT and [F 18]FDG PET/CT scans for his/her cancer care
* Patient must have hepatic and renal functions as defined by laboratory results within the following ranges:

  * Total bilirubin within 2 times institutional upper limit of normal
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 times institutional upper limits of normal
  * Serum creatinine ≤ 2.5 times institutional limit of normal
  * BUN within 2 times institutional upper limit of normal

Exclusion Criteria:

* Patient is not capable of complying with study procedures
* Female patient is pregnant or nursing

  o Exclude the possibility of pregnancy by one of the following:
  * Confirming in medical history that the patient is post-menopausal for a minimum of one year, or surgically sterile
  * Confirming the patient is using one of the following methods of birth control for a minimum of one month prior to entry into this study: IUD, oral contraceptives, Depo-Provera, or Norplant
  * Confirming a negative urine dipstick test taken the morning of but before receiving [F 18]HX4
* Patient has been involved in an investigative, radioactive research procedure within 7 days and during the study participation period
* Patient has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Brunetti, MD, Principal Investigator — Holy Name Hospital; Orhan Nalcioglu, PhD, Principal Investigator — University of California Irvine Medical Center, Orange, CA; Alan Waxman, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, CA; Kyung-Han Lee, MD, Principal Investigator — Sungkyunkwan University School of Medicine, Samsung Medical Center, Gangnam-gu, Seoul, Korea; Dae-Hyuk Moon, MD, Principal Investigator — University of Ulsan College of Medicine, Asan Medical Center, Songpa-gu, Seoul, Korea; Scott Dessain, MD, PhD, Principal Investigator — Lankenau Institute for Medical Research, Wynnewood, PA and Bryn Mawr Hospital Outpatient Imaging Center, Bryn Mawr, PA; Rathan Subamaniam, MD, Principal Investigator — Boston Medical Center, Boston, MA; Shyam Srinivas, MD, PhD, Principal Investigator — Cleveland Clinic, Cleveland, OH; Nasrin Ghesani, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey, NJMS-UH/UMDNJ Cancer Center, and University Heights Advanced Imaging Center, Newark, NJ; John M Buatti, MD, Principal Investigator — University of Iowa Hospitals and Clinics, Carver College of Medicine, and Holden Comprehensive Cancer Center,Iowa City, Iowa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 patients were enrolled into the study. There were 42 of 50 patients received at least one dose of [F-18]HX4 and had safety data collected. There were 39 of 50 patients completed two pre-treatment [F-18]HX4 PET/CT scans and were included in analyses to assess reproducibility.
Groups:
- [F 18]HX4: [F 18]HX4 : Approximately forty (40) patients who have diagnosis confirmed by histopathological examination of tumor tissue from head/neck, lung, liver, rectal or cervical cancers and will receive chemotherapy, radiation therapy or chemoradiotherapy, will be imaged under PET/CT with [F 18]HX4
Period: Overall Study
Arm/Group | [F 18]HX4
Started | 50 (A total of 50 patients were enrolled into the study.)
Completed | 42 (42 of 50 patients received at least one dose and 39 of 50 patients completed two pre-treatment scan)
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: A total of 50 patients were enrolled. A total of 42 patients received at least one dose of [F-18]HX4. Thirty-nine (39) patients completed two pre-treatment [F-18]HX4 PET/CT scans. Thirty (30) patients had an evaluable tumor response assessment 3 (±1) months after treatment start
Arm/Group | [F 18]HX4
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 10
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Reproducibility of [F18]HX4 PET Imaging in Measuring Hypoxia in Tumors
Description: Primary tumor uptake of [F 18]HX4 was measured on PET images by onsite radiologist or nuclear medicine physician for 1st and 2nd PET scans. Values measured were: SUV (Standard Uptake Value), SUV Max (Maximum standard uptake value), SUV Mean (Mean standard uptake value), and T/B ratio (Tumor to background ratio). Pearson's correlation coefficient was calculated for each of the parameter.
Time Frame: Time between 1st and 2nd scan was 1 to 6 days
Population: Based upon inclusion/exclusion criteria
Measure: Number; unit: participants
Groups:
- Subjects That Received 1st and 2nd [F18] HX4 Scans: Single arm study. This group includes all subjects that successfully received [F18]HX4 PET scan on 2 separate occasions within 6 days apart to assess reproducibility in measuring tumor hypoxia.
Arm/Group | Subjects That Received 1st and 2nd [F18] HX4 Scans
Number analyzed (Participants) | 39
participants | 39
Statistical Analysis 1: Comparison: Subjects That Received 1st and 2nd [F18] HX4 Scans; Primary Tumor SUV max: The reproducibility of [F-18]HX4 uptake in primary tumors was assessed by comparing SUV max of the 1st and 2nd [F18]HX4 PET/CT scan. Estimated power for a range of coefficients of variation (CVs) postulated for the paired differences in SUV values, and for establishing reproducibility within ±20% or ±25%; Test type: Superiority or Other; p < 0.001, Pearson's correlation — Significance of probability for no association between the first and second pre-treatment uptake; Pearson's Correlation Coefficient = 0.883, 90% CI 2-sided [0.802 to 0.929]
Statistical Analysis 2: Comparison: Subjects That Received 1st and 2nd [F18] HX4 Scans; Primary Tumor SUV mean: The reproducibility of [F-18]HX4 uptake in primary tumors was assessed by comparing SUV mean of the 1st and 2nd [F18]HX4 PET/CT scan. Estimated power for a range of coefficients of variation (CVs) postulated for the paired differences in SUV values, and for establishing reproducibility within ±20% or ±25%; Test type: Superiority or Other; p < 0.001, Pearson's correlation — Significance of probability for no association between the first and second pre-treatment uptake; Pearson's Correlation Coefficient = 0.887, 90% CI 2-sided [0.792 to 0.925]
Statistical Analysis 3: Comparison: Subjects That Received 1st and 2nd [F18] HX4 Scans; Primary Tumor to background SUV ratio: The reproducibility of [F-18]HX4 uptake in primary tumors was assessed by comparing tumor to background SUV ratio (T/B) of the 1st and 2nd [F18]HX4 PET/CT scan. Estimated power for a range of coefficients of variation (CVs) postulated for the paired differences in T/B values, and for establishing reproducibility within ±20% or ±25%; Test type: Superiority or Other; p < 0.001, Pearson's correlation — Significance of probability for no association between the first and second pre-treatment uptake; Pearson's Correlation Coefficient = 0.945, 90% CI 2-sided [0.904 to 0.967]

ADVERSE EVENTS:
Arm/Group | [F 18]HX4
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No